CLINICAL TRIAL: NCT05684042
Title: Fracture Database of the University Hospital Basel: A REDCap Assisted Reliability and Validity Study of Fracture Classifications of the Distal Radius
Brief Title: Fracture Registry University Hospital Basel
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-00921; mu22Bilici
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Distal Radius Fracture
Keywords: Fracture Database; Fracture Classifications of the Distal Radius; Quality assurance; REDCap
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data analysis: Accuracy measurement of the classifications of the distal radius fracture in the fracture database. — An expert panel (3 in-house experienced specialists) carries out a new fracture classification based on the anonymous radiological images in the interface of the REDCap fracture database. The degree of discrepancy between the expert panel and the database in fracture classifications is analyzed. By evaluating the extracted data, it is analyzed how valid the quality of the collected fracture classifications are, which the medical staff carry out in everyday clinical practice.

SUMMARY:
The primary goal of this research project is to measure the accuracy of the classifications of the distal radius fracture in the fracture database. The evaluation of the extracted data analyzes the validity of the fracture classifications that the medical staff carry out in everyday clinical practice.

Endpoint of this project is the reclassification of the selected fractures by an in-house group of experts in order to be able to carry out a subsequent statistical evaluation. It is analyzed whether there are significant deviations between the classifications of the expert group and the fracture database.

DETAILED DESCRIPTION:
Since 2017, a fracture database has been developed in the Department of Orthopedics and Traumatology at the University Hospital in Basel. Since November 2018, all patients who are treated surgically in the Clinic for Traumatology & Orthopedics due to fractures of the extremities or the pelvis have been included in the fracture database of the University Hospital Basel for quality assurance purposes.

This database was created with the research software REDCap and is used for internal quality measurement. It essentially consists of three instruments: the encoded patient data, the diagnosis and the therapy. In order to promote rapid digitized progress in the health care system, the quality of the recorded data must be checked regularly through suitable studies. This type of quality management is of essential scientific relevance for the fracture database of the University Hospital Basel. For this reason, the classifications of the recorded fractures in the database are to be examined on a random basis so that weak points in the system can be addressed and staff can be better trained. The primary goal of the project is to measure the accuracy of the classifications of the distal radius fracture in the fracture database. The evaluation of the extracted data analyzes the validity of the fracture classifications that the medical staff carry out in everyday clinical practice.

Endpoint of this project is the reclassification of the selected fractures by an in-house group of experts in order to be able to carry out a subsequent statistical evaluation. It is analyzed whether there are significant deviations between the classifications of the expert group and the fracture database.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 16 years of age and regardless of gender
* Surgical treatment of a primary fracture of the distal radius was performed
* Pre-therapeutic radiographs of good quality and in two planes
* General consent for quality assurance and research was not rejected

Exclusion Criteria:

* Existence of a documented refusal
* Patients under the age of 16, as they are treated in the children's hospital
* Conservative treatment of the distal radius fracture
* Re-fracture after conservative or surgical treatment
* Incorrect planes and poor quality of X-rays
* Exclusive performance of a computed tomography, e.g. after polytrauma
* Duplicates within the database
* X-rays with forearm cast

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The health-related and personal data and all image material (X-rays) come from patients who were treated for surgical treatment of a distal radius fracture in the Clinic for Traumatology & Orthopedics at the University Hospital Basel. The REDCap database has been a tool for quality assurance in patient care at the USB since November 2018. The medical staff records all relevant data on a daily basis and archives it under data protection guidelines.
Sampling Method: Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2033-06 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Number of discrepancies between the classifications of the expert group and the fracture database | one time assessment at baseline
  Number of discrepancies between the classifications of the expert group and the fracture database

CONTACTS AND LOCATIONS:
Overall Officials: Murat Bilici, Principal Investigator — University Hospital Basel, Clinic for Orthopedics and Traumatology
Locations (1):
- University Hospital Basel, Orthopedics and Traumatology, Basel, Switzerland